CLINICAL TRIAL: NCT05517200
Title: Pilot Study for Machine Learning as Applied to EEG as an Aid to the Diagnosis of Adult Migraineurs Without Aura, or Migraineurs With Aura on Interictal (Non-pain) Days
Brief Title: Pilot Study for a Machine Learning Test for Migraine
Acronym: MLTM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Headache Sciences Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: MLTM1
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Migraine; Chronic Migraine; Tension-Type Headache
Keywords: EEG; Machine Learning; Migraine; Headache; Diagnosis; Artificial Intelligence
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Headache; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Control: These participants are normal control in good mental and psychiatric health.
  Interventions: Diagnostic Test: Machine Learning Test for Migraine
- Migraine: These participants have migraines according to ICHD-3 criteria.
  Interventions: Diagnostic Test: Machine Learning Test for Migraine

INTERVENTIONS:
Diagnostic Test: Machine Learning Test for Migraine — Resting EEG, and Visual and Auditory Stimulation
  Other Names: MLTM

SUMMARY:
This study is a single center, random participant selection, data analyst is blinded to patient identifiers, controlled clinical trial.

The proposed study is intended to establish safety and efficacy of quantifiable electrical biomarkers for migraine that can be used to confirm a diagnosis in people that have already been screened as positive for migraine using the gold standard participative criteria set out in the International Classification of Headache disorders-3 (ICHD-3) criteria.

It is hypothesized that specific brain signals can be used to distinguish between migraine patients with and without aura from normal control and tension- type headache control participants by EEG enhanced with machine learning software.

ELIGIBILITY:
Inclusion Criteria:

* ● Age range: All participants and controls will be adults over 18, and no greater than 70

  * Sex: Migraine patients and controls to reflect the demographics of the disease such that there is a balanced mix of males to females that reflects known female to male ratio for migraine is 3 to 1.
  * Capable of giving clear and reliable answers on the questionnaires
  * All potential participants should be able to read, write and speak in English: unless they can bring a translator.
  * All mentally competent: to give accurate answers on questionnaires, to decide for themselves and sign the informed consent form.
  * All medically stable patients.
  * Capable of safely using a staircase to our downstairs lab
  * OHIP must be up-to-date and participants must show a valid OHIP number
  * Able and willing to comply with all study requirements
  * Normal controls must be very healthy.

Exclusion Criteria:

* ● Under 18 years old

  * Over 70 years old (71 and above)
  * Incompetent in english language and no translator (This applies to reading, writing and speaking.)
  * Current moderate or serious mental illness (including depression, anxiety disorder, psychosis)
  * Mentally disabled/ Mentally incompetentHistory of photo-epilepsy or history of seizure following shortly after visual stimulus such as bright or repetitive flashes of light, repetitive flashes of light (such as at a disco, or looking at an overhead fan), or after looking at repetitive visual patterns lines such as looking at multiple stripes or squares, or from seeing movement such as when watching an action movie.
  * Medically unstable
  * Prisoner
  * Unable to go down the stairs (if recording is downstairs)
  * Pacemaker
  * Defibrillator
  * Cochlear implants
  * Significant skull deformity (e.g. a depression of greater than half an inch
  * Head injury with consciousness loss in the last year, even with apparent full recovery.
  * Severe facial trauma within the last three months, or longer if unrecovered.
  * Unnatural material inside the head or mouth based on history (including clips from surgery, shrapnel, bullet, medical pump, wires, medical device, metal dental implants)
  * Chronic communicable diseases carried (including Hepatitis B, Hepatitis C, HIV, Creutzfeldt-Jakob Disease) Note: Vagal stimulator and insulin pump are not an exclusion criteria, but must be turned off before the EEG recording starts.

4.2.2 EXCLUSION CRITERIA FOR NORMAL CONTROLS

* not in excellent physical health
* not in excellent neurological health and especially, no headache disorder at all in the last three months
* not in excellent mental health
* no central sensitization disorder (For details see section for "Central Sensitization Questionnaires" in the document called "General Headache Registration and History Form For Migraine With Aura, Migraine Without Aura and Normal Controls and Frequent Tension-Type Headache Controls". (See documents provided to Veritas IRB via Concierge.)
* not a good sleeper
* no chronic pain disorder
* No psychoactive drugs for 2 weeks before recording day
* Not currently in pain on recording day
* No neurological illness
* No known moderate to severe mental illness 4.2.3 EXCLUSION CRITERIA FOR MIGRAINE WITH AURA:
* Chronic migraine with aura

4.2.3 EXCLUSION CRITERIA FOR MIGRAINE WITHOUT AURA:

● Chronic migraine without aura

4.2.4 EXCLUSION CRITERIA FOR TENSION-TYPE HEADACHES:

* A history of migraine (including any presently suspected to have recent migraine)
* Chronic tension-type headache

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants and controls will be adults over 18, and no greater than 70. Migraine patients and controls to reflect the demographics of the disease such that there is a balanced mix of males to females that reflects known female to male ratio for migraine is 3 to 1. They are capable of giving clear and reliable answers on the questionnaires. All potential participants should be able to read, write and speak in English, unless they can bring a translator. All mentally competent to give accurate answers on questionnaires, to decide for themselves and sign the informed consent form. All medically stable patients. Capable of safely using a staircase to our downstairs lab. Normal controls must be very healthy.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of machine learning as applied to EEG to diagnose migraine. | 2 years
  The primary endpoint is a sensitivity of 79% and a specificity of 72% in distinguishing migraine with and without aura screened using the ICHD-3 benchmark criteria as compared to normal controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Sciences Incorporated Laboratory, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: United States ( 12 ) Patent Application Publication Pub . No . : US 2018 / 0242919 A1 DOIDGE et al . ( 43 ) Pub . Date : Aug . 30 , 2018 ( 54 ) DIAGNOSIS OF MIGRAINE VIA EXPERT SYSTEM — https://patentimages.storage.googleapis.com/df/b6/d0/d21792f1e6cdd0/US20180242919A1.pdf